CLINICAL TRIAL: NCT03323138
Title: Prospective Study on Ex-PRESS Implantation Combined With Phacoemulsification in Primary Angle-closure Glaucoma
Brief Title: Study on Ex-PRESS Implantation Combined With Phacoemulsification in Primary Angle-closure Glaucoma
Acronym: PACG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, MD, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL-HZ
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Glaucoma, Angle-Closure
Keywords: Ex-PRESS; glaucoma; filtration surgery; phacoemulsification
MeSH Terms: conditions — Glaucoma, Angle-Closure; Glaucoma | interventions — Phacoemulsification

STUDY DESIGN:
Intervention Model Description: Prospective, interventional and monocentric study based in a university hospital setting
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ex-PRESS and phacoemulsification (Experimental): A treatment session of PACG coexisting cataract treated with phacoemulsification combined with P50 Ex-PRESS miniature glaucoma device (Alcon Laboratories, Fort Worth, Texas, USA).
  Interventions: Procedure: Ex-PRESS and phacoemulsification

INTERVENTIONS:
Procedure: Ex-PRESS and phacoemulsification

SUMMARY:
Primary angle-closure glaucoma (PACG) is common, phacotrabeculectomy is associated with a significant risk of complications.The Ex-PRESS shunt was introduced as a modification to trabeculectomy, with the theoretical advantages of reduced complications.Our purpose is to perform a prospective study to evaluate the clinical outcomes and safety of the Ex-PRESS shunt with cataract surgery for PACG patients coexisting cataract.

DETAILED DESCRIPTION:
The Ex-PRESS is a miniature stainless steel glaucoma device, developed as an alternative to trabeculectomy mainly for patients with primary open-angle glaucoma.It has been proved to be as effective as trabeculectomy in a series of researches. However the early postoperative complication of Ex-PRESS implantation is less frequent compared with trabeculectomy. Ex-PRESS was designed initially for open angle glaucoma, gradually some scholars used it in refractory postpenetrating keratoplasty glaucoma and in vitrectomized glaucoma,which showed that Ex-PRESS shunt implantation was an effective procedure too. We analyzed the clinical efficacy and safety of combined phacoemulsification and Ex-PRESS implantation for PACG patients with cataract. Data was recorded before surgery and postoperatively at 1 week and 1, 3, 6, 12,18,24,30,36 months，which included intraocular pressure (IOP), best corrected visual acuity (BCVA), number of medications, complications, corneal endothelial cell density and anterior segment optical coherence tomography(AS-OCT). Efficacy was assessed by IOP values and success rates. Complete success was determined by IOP between 5 and 21mmHg without medications.

ELIGIBILITY:
Inclusion Criteria:

* The presence of PACG, angle peripheral anterior synechia (PAS) more than 180 degrees.
* An indication for glaucoma filtering surgery based on uncontrolled IOP or progressive vision field defect despite antiglaucoma medications.
* Mean vision field defect greater than 15dB.
* The presence of a clinically significant decrease of visual acuity as a result of cataract, usually BCVA less than 0.6.

Exclusion Criteria:

* Patients unable to give informed consent.
* Ocular infection or inflammation in the study eye in the 3 months prior to enrollment.
* Intraocular surgery in the study eye in the 3 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | 36 months
  In millimeters of mercury (mmHg), measured with the Goldmann applanation tonometer

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | 2 weeks, 1 month, 3 months, 6 months, 12 months,18 months, 24 months, 30 months,36 months.
  In millimeters of mercury (mmHg), measured with the Goldmann applanation tonometer
Number of intraocular pressure lowering medications | 2 weeks, 1 month, 3 months, 6 months, 12 months,18 months, 24 months, 30 months,36 months.
  Number of drops and oral medications used by the patient compared to baseline
Best corrected visual acuity (BCVA) | 2 weeks, 1 month, 3 months, 6 months, 12 months,18 months, 24 months, 30 months,36 months.
  Number of lines reduction or improvement from baseline on Snellen acuity chart
Corneal endothelial cell density | 3 months
  Use non-contact specular microscope to count the endothelial cell density (cells/mm2)
Anterior chamber distance(ACD) | 3 months
  The distance from inner corneal surface to lens measured by AS-OCT
Angle opening distance(AOD500) | 3 months
  Angle opening distance 500um from the scleral spur measured by AS-OCT

CONTACTS AND LOCATIONS:
Overall Officials: Ai wu Fang, MD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Ophthalmology and Optometry Hospital , Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lai JS, Tham CC, Lam DS. Incisional surgery for angle closure glaucoma. Semin Ophthalmol. 2002 Jun;17(2):92-9. doi: 10.1076/soph.17.2.92.14716. PMID 15513462
- [Result] Tham CC, Lai JS, Poon AS, Lai TY, Lam DS. Results of trabeculectomy with adjunctive intraoperative mitomycin C in Chinese patients with glaucoma. Ophthalmic Surg Lasers Imaging. 2006 Jan-Feb;37(1):33-41. PMID 16468549
- [Result] Tham CC, Kwong YY, Leung DY, Lam SW, Li FC, Chiu TY, Chan JC, Lam DS, Lai JS. Phacoemulsification versus combined phacotrabeculectomy in medically uncontrolled chronic angle closure glaucoma with cataracts. Ophthalmology. 2009 Apr;116(4):725-31, 731.e1-3. doi: 10.1016/j.ophtha.2008.12.054. Epub 2009 Feb 25. PMID 19243831
- [Result] Beltran-Agullo L, Trope GE, Jin Y, Wagschal LD, Jinapriya D, Buys YM. Comparison of visual recovery following ex-PRESS versus trabeculectomy: results of a prospective randomized controlled trial. J Glaucoma. 2015 Mar;24(3):181-6. doi: 10.1097/IJG.0b013e31829e1b68. PMID 23807352
- [Result] Gonzalez-Rodriguez JM, Trope GE, Drori-Wagschal L, Jinapriya D, Buys YM. Comparison of trabeculectomy versus Ex-PRESS: 3-year follow-up. Br J Ophthalmol. 2016 Sep;100(9):1269-73. doi: 10.1136/bjophthalmol-2015-307161. Epub 2015 Dec 16. PMID 26674779
- [Result] Netland PA, Sarkisian SR Jr, Moster MR, Ahmed II, Condon G, Salim S, Sherwood MB, Siegfried CJ. Randomized, prospective, comparative trial of EX-PRESS glaucoma filtration device versus trabeculectomy (XVT study). Am J Ophthalmol. 2014 Feb;157(2):433-440.e3. doi: 10.1016/j.ajo.2013.09.014. Epub 2013 Nov 7. PMID 24210765
- [Result] Zhang M, Li B, Sun Y. EX-PRESS and ahmed glaucoma valve in treatment of refractory glaucoma. Acta Ophthalmol. 2016 Aug;94(5):e382-3. doi: 10.1111/aos.12898. Epub 2015 Dec 8. No abstract available. PMID 26643962
- [Result] Liu B, Guo DD, Du XJ, Cong CY, Ma XH. Evaluation of Ex-PRESS implantation combined with phacoemulsification in primary angle-closure glaucoma. Medicine (Baltimore). 2016 Sep;95(36):e4613. doi: 10.1097/MD.0000000000004613. PMID 27603352
- [Result] Wagschal LD, Trope GE, Jinapriya D, Jin YP, Buys YM. Prospective Randomized Study Comparing Ex-PRESS to Trabeculectomy: 1-Year Results. J Glaucoma. 2015 Oct-Nov;24(8):624-9. doi: 10.1097/IJG.0000000000000029. PMID 24247999
- [Result] Marzette L, Herndon LW. A comparison of the Ex-PRESS mini glaucoma shunt with standard trabeculectomy in the surgical treatment of glaucoma. Ophthalmic Surg Lasers Imaging. 2011 Nov-Dec;42(6):453-9. doi: 10.3928/15428877-20111017-03. PMID 22074705
- [Result] Vetrugno M, Ferreri P, Sborgia C. Ex-PRESS miniature glaucoma device in vitrectomized eyes. Eur J Ophthalmol. 2010 Sep-Oct;20(5):945-7. doi: 10.1177/112067211002000521. PMID 20306441
- [Result] Kanner EM, Netland PA, Sarkisian SR Jr, Du H. Ex-PRESS miniature glaucoma device implanted under a scleral flap alone or combined with phacoemulsification cataract surgery. J Glaucoma. 2009 Aug;18(6):488-91. doi: 10.1097/IJG.0b013e31818fb44e. PMID 19223790